CLINICAL TRIAL: NCT06420011
Title: A Real-World, Observational, Multicentre Retrospective Analysis to Evaluate the Clinical Characteristics, Medical Management and Outcomes of Hospitalised Patients With Factor XA Inhibitor-Related InTracranial Haemorrhage (FAITH)
Brief Title: FAITH - Factor XA Inhibitor-Related InTracranial Haemorrhage
Acronym: FAITH
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D9603R00022
Record Dates: First submitted 2024-03-04; First posted 2024-05-17 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-08

CONDITIONS: InTracranial Haemorrhage
Keywords: Factor XA Inhibitor-Related InTracranial Haemorrhage; FXa; ICH; FAITH
MeSH Terms: conditions — Intracranial Hemorrhages

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
FAITH study is a multicentre retrospective analysis study that aims to understand the burden of ICH related to FXa inhibitors and the current treatment approaches in country/countries where specific reversal agents are not available yet. The results of this analysis will improve our understanding of FXa inhibitor-related ICH, its socioeconomic impact and factors associated with negative outcomes in real-world settings. The insights gained can inform clinical decision making and potentially lead to strategies to optimise the use of FXa inhibitors, increase the availability of specific reversal agents and improve patient safety and outcomes.

DETAILED DESCRIPTION:
FAITH is a retrospective, non-interventional, multicentre cohort study that will retrieve the data from medical records of adult patients who were hospitalised with confirmed diagnosis of ICH while being treated with FXa inhibitors. The primary objectives of the study is to describe the characteristics and hospital outcomes of hospitalised patients with FXa inhibitors-related ICH in real-world settings. Data of consecutive patients admitted on or after 1 January 2021 and by 30 June 2023 will be retrieved. The index date is defined as the date of hospital admission.The identification of ICH will be based on the CT/MRI scan records and according to the ICD-10-CM diagnosis code. To establish the causal relation between FXa and ICH, the study will include only patients who were determined in the medical records to have taken oral FXa inhibitors.The historical data will be followed up from the index date (the date of hospital admission) until the earliest date of death, lost to follow-up or up to 6 months.The 6-month follow-up period will allow for the assessment of the disability rate and the need for supportive care among survivors.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥ 18 years of age at the time of hospital admission.
* Patients presented with a spontaneous or traumatic haemorrhage into any intracranial compartment. The diagnosis of ICH will be based on Computed Tomography (CT) or Magnetic Resonance Imaging (MRI) scan and according to the ICD-10-CM diagnosis code.
* Patients who were determined in the medical records to have taken a dose of oral FXa inhibitors within 24 hrs before hospital presentation that warranted reversal of anticoagulant activities.

Exclusion Criteria:

* Patients who were treated with andexanet alfa.
* Patients who were enrolled in any clinical trials during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will recruit 350 adult patients (age ≥18 years at the time of hospital admission) hospitalised patients with FXa inhibitors-related ICH from a total of 20-25 sites from Asia-Pacific Region, Latin America, and the MEA, where FXa inhibitors specific reversal agent is not approved locally.
Sampling Method: Non-Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2024-07-08 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Patient characteristics | Index day (Date of hospitalization) to 24hours
  Age of the patients at the time of hospital admission (years) is recorded on Index day within 24 hours of hospitalization
Patient Characteristics | Index day (Date of hospitalization) to 24hours
  Race (Middle Eastern, Asian, other) of the eligible patients is collected
Sociodemographic Characteristics of eligible patients | Index day (Date of hospitalization) to 24hours
  Sociodemographic characteristics like Sex (Male or Female) of the eligible patients is recorded on Index day
Sociodemographic Characteristics | Index day (Date of hospitalization) to 24hours
  Sociodemographic characteristics like nationality of the eligible patients info is collected on Index day
Clinical characteristics | Index day (Date of hospitalization) to 24hours
  Comorbidities info of the eligible patients is recorded on Index day
Clinical Characteristics | Index day (Date of hospitalization) to 24hours
  Clinical characteristics like BMI in Kg/m2 of the eligible patients is recorded on Index day
FXa inhibitor characteristics | Time of last Fxa inhibitor dose to the time of hospital admission of maximum 24 hours
  At index date the following FXa inhibitor characteristics will be described :
  Indication ,type and dose pf FXa Inhibitor
ICH characteristics | Index day to 1 week
  The primary ICH characteristics like type, site and presence of multicompartment haemorrhage during hospitalisation from Index date to 24hours
GCS score | Index day to 24hours
  The GCS is scored between 3 and 15. 3 being the worst and 15 the best. It is composed of three parameters: best eye response (E), best verbal response (V), and best motor response (M)
mRS score | Index day to 24 hours
  mRS score recorded within 24 hours on Index date The mRS is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or others causes of neurological disability. It is scored from: 0=No symptoms at all
  1. No significant disability
  2. Slight disability
  3. Moderate disability
  4. Moderately severe disability 5=Severe disability
  6=death
NIHSS score | Index date up to 24 hours
  NIHSS score recorded within 24 hours on the Index date
  Scores range from 0 to 42, with higher scores indicating greater severity. Stroke severity may be stratified on the basis of NIHSS scores as follows:
  Very Severe: >25 Severe: 15 - 24 Mild to Moderately Severe: 5 - 14 Mild: 1 - 5
Haematoma volume | Index day to 24 hours
  Haematoma volume based on baseline Imaging scans taken within 24 hours on the index date
BP (Systolic and Diastolic) | Index day to 72 hours
  BP at Index date during hospital admission and in 6, 24, and 72 hours
Antihypertensive treatment | Index day to 1 Week
  Antihypertensive treatment patterns during hospitalisation from Index date to 1 week
In-hospital mortality due to any cause | Index date up to the death event during hospital stay (maximum 1 week)
  Number of patients died between index date (date of hospitalization) to Hospital discharge (maximum of 1 week)
Mortality at 30 days, post index event | Index date up to 30 days
  Number of patients died between index date (date of hospitalization) up to 30 days
Mortality at 3 months post index event | Index date up to 3 months
  Number of patients died between index date (date of hospitalization) up to 3 months
Mortality at 6 months post index event | Index date up to 6 months
  Number of patients died between index date (date of hospitalization) up to 6 months
Type of discharge disposition | Hospital discharge to Maximum of 6 months
  During the period from the hospital discharge date up to death event or 6 months, whichever occurs first, the following type of hospital discharge disposition will be described for survivors like Home, inpatient rehabilitation facility, nursing home, other hospitals/medical centres

SECONDARY OUTCOMES:
Time from symptoms onset to hospital admission | Baseline (which is the date of hospitalization i.e. Index date) to a maximum of 24 hours
  Time between the onset of the bleeding symptoms to admission of patient in hospital in hours.
Time from Hospital admission to time taken to do Imaging scan | Index day (Date of hospitalization) to Maximum of one hour
  Time between patient hospital admission to the performing of Imaging scan in minutes, less than 1 hour
Time from hospital admission to administration of any haemostatic therapy | Index day (Date of hospitalization) to Maximum of one hour
  Time between patient hospital admission to start of the any haemostatic therapy in minutes, in less than 1 hour
Healthcare resource utilization during hospitalisation | Index day to maximum of 1 week
  The length of ICU stay of eligible patients in days from Index day to maximum of 1 week
Length of hospitalisation in days | Index day to maximum of 1 week
  The length of hospitalisation of eligible patients in days from Index day to maximum of 1 week
Disability rate among survivors | At hospital discharge (Maximum of 1 week from Index day)
  At hospital discharge (Maximum of 1 week from Index day) Modified Rankin Score (mRS) will be described
  Functional outcome assessed with the modified Rankin Scale (mRS) at hospital discharge .The mRS is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered of stroke or other causes of neurological disability. It is scored from:
  0=No symptoms at all
  1=No significant disability, 2=Slight disability 3=Moderate disability 4=Moderately severe disability 5=Severe disability 6=death
Disability rate among survivors | Index day to 3 months
  At three months, after the index event (date of hospital admission) Modified Rankin Score (mRS) will be described.
Health care resource utilization after hospital admission up to 6 months | Index date to 6 months
  From the index date to 6 months the following HCRU will be described:
  Need for supportive medical care ,type of supportive care (including rehabilitation services), inpatient rehabilitation, outpatient rehabilitation, including occupational therapists, speech and language pathologists, dietician, nurse, adaptive equipment, everything else.
Health care resource utilization within 6 months after hospital discharge. | Hospital discharge up to 6 months
  From the patient hospital discharge up to 6 months the following HCRU will be described:
  Number of inpatient readmissions after discharge and up to 6 months, Type of ward, Number of days of hospitalization Reason for readmission and Medications.
Disability rate among survivors | Index day to Maximum of 6 months
  At six months after the index event (date of hospital admission) Modified Rankin Score (mRS) will be described.

CONTACTS AND LOCATIONS:
Locations (10):
- Research Site, Buenos Aires, Argentina
- Brazil (2):
  - Research Site, Joinville
  - Research Site, Porto Alegre
- Research Site, Bogotá, Colombia
- Research Site, Mexico City, Mexico
- Research Site, Doha, Qatar
- Saudi Arabia (2):
  - Research Site, Mecca
  - Research Site, Riyadh
- United Arab Emirates (2):
  - Research Site, Abu Dhabi
  - Research Site, Al Ain City

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Redacted CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9603R00022&attachmentIdentifier=2e131dfe-29f5-4a16-82cc-25475dd74215&fileName=D9603R00022_Redacted_CSR_synopsis.pdf&versionIdentifier=